CLINICAL TRIAL: NCT05267080
Title: Registry on Percutaneous Electrochemotherapy
Acronym: RESPECT
Status: Active, not recruiting | Type: Observational
Sponsor: Cardiovascular and Interventional Radiological Society of Europe (Other)
Responsible Party: Sponsor
Other Study IDs: RESPECT
Record Dates: First submitted 2022-02-11; First posted 2022-03-04 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Primary Liver Cancer; Secondary Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: CLINIPORATOR — The CLINIPORATOR is used to perform percutaneous electrochemotherapy on liver tumours.

SUMMARY:
The Registry on Percutaneous ElectroChemoTherapy (RESPECT) is a post-market, prospective, non-randomized, observational study aiming at evaluating the effectiveness of percutaneous electrochemotherapy (ECT) for the treatment of liver cancer.

DETAILED DESCRIPTION:
Electrochemotherapy (ECT) is a local tumour ablation technique that uses reversible electroporation to transiently permeabilize the cell membrane in order to increase the cytotoxicity of chemotherapeutic drugs. A major advantage of ECT is that its antitumour efficacy is driven by the chemotherapeutic agent which predominantly targets rapidly-dividing tumour cells, with very little collateral damage on neighbouring structures.

ECT is typically performed using the CLINIPORATOR®, a medical grade pulse generator for clinical electroporation, whose development was funded by the European Commission in an effort to standardize the operating procedures for ECT. The feasibility, safety and efficacy of ECT with the CLINIPORATOR® have been consistently reported for the management of different types of primary and secondary liver cancers: colorectal liver metastasis, hepatocellular carcinoma, portal vein tumour thrombosis from hepatocellular carcinoma, perihilar cholangiocarcinoma and liver metastasis from renal cancer.

While ECT for liver malignancies has been mostly performed intraoperatively, recent studies have successfully used a percutaneous approach. These studies, which were either single-case reports or involved a very limited number of patients (< 10), have introduced percutaneous ECT as a very promising minimally invasive treatment option for liver cancer, with the obvious benefits of fewer surgical complications, faster recovery and shorter hospitalization. However, results from a larger and more diverse patient population are needed in order to confirm its therapeutic efficacy.

The aim of the RESPECT study is to expand our understanding of percutaneous ECT for primary and secondary liver cancer by 1) substantiating the evidence base for the effectiveness and safety of percutaneous ECT in a large-scale, multi-centric, cross-border sample; and 2) extending the current evidence base regarding percutaneous ECT with appropriately defined follow-up data, as well as information regarding quality of life.

RESPECT is a post-market, prospective, non-randomized, observational study. Patients with any type of liver cancer will be given the possibility to enrol after they are referred to percutaneous ECT by a multidisciplinary tumour board, hence participation to the registry neither affects treatment plan nor influence treatment quality. Patient enrolment will last 3 years, with a follow-up period of 1 year. Data will be collected less than 1 week before treatment (baseline) and at different intervals following treatment (1 day, 2 weeks, 1 month, 3 months, 6 months, 12 months, and every 6 months until the end of the study). Effectiveness of ECT will be primarily assessed by the status of each treated lesion 12 months after treatment. Overall survival, overall local disease-free survival, hepatic disease-free survival, time to untreatable progression by ECT and vacation from systemic cancer therapy will give further insight into the impact of ECT. Safety will be evaluated based on the occurrence and severity of adverse events associated with the treatment. Quality of life and pain will be documented using questionnaires filled by the patients at the first 3 to 4 follow-ups.

Overall, RESPECT intends to provide healthcare professionals and health authorities with information on percutaneous ECT for liver cancer to help decision-making regarding treatment access and treatment modalities and optimize patient care.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Primary or secondary liver cancer
* Referral to local ablative treatment by multidisciplinary tumour board and decision to treat with pECT by interventional radiologist in charge
* Planned treatment with pECT using the CLINIPORATOR
* Signed informed consent form

Exclusion Criteria:

Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary or secondary liver cancer referred to local ablative treatment by multidisciplinary tumour board and treated with pECT by decision of the interventional radiologist in charge.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2026-01-23 (Actual); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Local Tumour Control | 12 months
  Based on the tumour status according to mRECIST assessment

SECONDARY OUTCOMES:
Safety (in terms of adverse events related to treatment) | 12 months
  Based on the occurrence of adverse events and their severity according to CTCAE v5.0
Tumour status (size) | End of study (maximum 36 months)
  Based on tumour size
Tumour status (mRECIST) | End of study (maximum 36 months)
  Based on mRECIST assessment
Quality of life (EORTC QLQ-C30) | 3 months
  Based on the Quality of Life questionnaire EORTC QLQ-C30 filled by the patients before ECT treatment and at different time intervals following ECT treatment.
  Quality of life data is measured according to three scales: functional scale, symptom scale and global health. On the functional scale, scores range from 1 to 4, with a score of 1 corresponding to no at all and a score of 4 corresponding to very much. On the symptom scale, scores range from 1 to 4, with a score of 1 corresponding to no at all and a score of 4 corresponding to very much.
  For global health, the scores range from 1 to 7, with a score of 1 corresponding to either very poor global health or very poor quality of life, and a score of 7 corresponding to either excellent global health or excellent quality of life.
Pain assessment | 1 month
  Based on the pain questionnaire filled by the patients before ECT treatment and at different time intervals following ECT treatment.
  Severity of pain is graded on a scale from 0 to 10, with 10 corresponding to the most severe pain. Pain frequency is graded from 0 (no pain) to 4 (chronic pain persistent for more than 3 months). Quality of pain is classified into 4 categories: no, somatic, visceral and neuropathic pain.
Effectiveness (Survival) | End of study (maximum 36 months)
  Survival will be categorized with respect to overall survival, overall local disease-free survival and hepatic disease-free survival
Effectiveness (Time to untreatable progression by ECT) | End of study (maximum 36 months)
  Based on the timeframe until the progressing tumour is not treatable by ECT anymore
Systemic cancer therapy vacation | End of study (maximum 36 months)
  Based on the time frame following ECT treatment during which patients do not need systemic cancer therapy
Economic aspects | 2 weeks
  Based on the duration of hospitalization following ECT treatment

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Wiggermann, Prof. Dr., Study Chair — Städtisches Klinikum Braunschweig, Braunschweig, Germany; Attila Kovács, PD. Dr. med., Study Chair — WEGE Klinik, Bonn, Germany; Franco Orsi, Prof., Study Chair — European Institute of Oncology, Milan, Italy
Locations (15):
- France (3):
  - Centre Hospitalier Universitaire de Montpellier, Montpellier
  - Hôpital Européen Georges-Pompidou, Paris
  - Institut Gustave Roussy, Paris
- Germany (5):
  - WEGE Klinik, Bonn
  - Städtisches Klinikum Braunschweig, Braunschweig
  - Universitätsklinikum Halle, Halle
  - Helios Park-Klinikum, Leipzig
  - University Hospital Regensburg, Regensburg
- University of Szeged, Szeged, Hungary
- Italy (3):
  - Istituto Europeo di Oncologia, Milan
  - Fondazione Policlinico Universitario Campus Bio-Medico, Rome
  - Policlinico Universitario A. Gemelli, Rome
- Vilnius University Hospital Santariškių Klinikos, Vilnius, Lithuania
- Hospital Universitario y Politécnico La Fe, Valencia, Spain
- Leeds Teaching Hospitals NHS Trust, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No